CLINICAL TRIAL: NCT00135382
Title: A Phase 3 Study Switching HIV-1 Infected Patients With an Undetectable Viral Load on a First Protease Inhibitor-Based Regimen to an Efavirenz-Based Regimen
Brief Title: Study Switching HIV-1 Infected Patients With an Undetectable Viral Load on a First Protease Inhibitor-Based Regimen to an Efavirenz-Based Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI266-406
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Didanosine; Lamivudine; efavirenz

INTERVENTIONS:
Drug: Videx EC
Drug: Epivir
Drug: Sustiva

SUMMARY:
The purpose of this study is to demonstrate that virologically controlled HIV-infected individuals can successfully switch from a protease inhibitor (PI)-based regimen to an efavirenz-based regimen while maintaining virologic control, as evaluated by the proportion of subjects who continue to have plasma HIV-1 levels < 50 copies/mL. In addition, a simplified once-daily regimen will improve adherence and quality of life.

DETAILED DESCRIPTION:
Patients randomized to the non Videx enteric coated (ddl EC)+lamivudine (3TC)+efavirenz (EFV) arm would continue their baseline nucleoside reverse transcriptase inhibitors (NRTIs) on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* ≥ 18 years of age and weight at least 40kg
* Two plasma HIV RNA levels < 50 copies/mL during the qualification and screening period
* Patients receiving a PI and ≥ 2 NRTIs

Exclusion Criteria:

* Pregnancy or breastfeeding
* Documented virologic failure while on their first PI-based antiretroviral (ARV) regimen
* Active AIDS-defining opportunistic infection or disease
* Proven or suspected acute hepatitis within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254
Dates: Start 2002-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Efficacy at week 48

SECONDARY OUTCOMES:
Safety, tolerability and efficacy at weeks (wks) 24 and 48; Effect on lipids at wks 24 and 48; Adherence, quality of life changes, treatment satisfaction and preference at wks 12, 24 and 48

CONTACTS AND LOCATIONS:
Locations (48):
- United States (46):
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Beverly Hills, California
  - Local Institution, Fountain Valley, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, San Diego, California
  - Local Institution, San Francisco, California
  - Local Institution, Tarzana, California
  - Local Institution, West Hollywood, California
  - Local Institution, Denver, Colorado
  - Local Institution, Norwalk, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Atlantis, Florida
  - Local Institution, Daytona Beach, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Miami Beach, Florida
  - Local Institution, North Miami, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Plantation, Florida
  - Local Institution, Safety Harbor, Florida
  - Local Institution, South Miami, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Decatur, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Boston, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, East Orange, New Jersey
  - Local Institution, Newark, New Jersey
  - Local Institution, Union, New Jersey
  - Local Institution, Brooklyn, New York
  - Local Institution, Manhasset, New York
  - Local Institution, Mount Vernon, New York
  - Local Institution, New York, New York
  - Local Institution, Stony Brook, New York
  - Local Institution, Valhalla, New York
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Hampton, Virginia
  - Local Institution, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Local Institution, Ponce
  - Local Institution, Rio Piedras